CLINICAL TRIAL: NCT02888691
Title: Low Carbohydrate Diet vs. High Carbohydrate Diet in Type 1 Diabetes: A Randomized Crossover Study
Brief Title: Low Carbohydrate Diet vs. High Carbohydrate Diet in Type 1 Diabetes
Acronym: HiLo12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Signe Schmidt, MD PhD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HiLo12
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): < 100 grams of carbohydrate per day
  Interventions: Other: Low carbohydrate diet
- High Carbohydrate Diet (Experimental): > 250 grams of carbohydrate per day
  Interventions: Other: High carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet
  Arms: Low Carbohydrate Diet
Other: High carbohydrate diet
  Arms: High Carbohydrate Diet

SUMMARY:
The aim of the study is to investigate glycemic control during a low carbohydrate diet compared with during a high carbohydrate diet in adults with insulin pump treated type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes ≥3 years
* Insulin pump use ≥1 year
* HbA1c ≥53 mmol/mol (7.0%)
* BMI 20-27 kg/m2
* Willingness to count carbohydrates and use the insulin pump bolus calculator for all boluses during the intervention periods
* Willingness to use continuous glucose monitoring consistently during the intervention periods

Exclusion Criteria:

* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Use of SGLT-2-inhibitors
* Use of corticosteroids during or within 30 days prior to the intervention periods
* Celiac disease
* Inflammatory bowel disease
* Macroalbuminuria
* Active proliferative retinopathy combined with an HbA1c ≥ 75 mmol/mol (9.0%)
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmidt S, Christensen MB, Serifovski N, Damm-Frydenberg C, Jensen JB, Floyel T, Storling J, Ranjan A, Norgaard K. Low versus high carbohydrate diet in type 1 diabetes: A 12-week randomized open-label crossover study. Diabetes Obes Metab. 2019 Jul;21(7):1680-1688. doi: 10.1111/dom.13725. Epub 2019 Apr 21. PMID 30924570
- [Derived] Ji L, Li L, Ma J, Li X, Li D, Meng B, Lu W, Sun J, Liu Y, Takayanagi G, Wang Y. Efficacy and safety of teneligliptin added to metformin in Chinese patients with type 2 diabetes mellitus inadequately controlled with metformin: A phase 3, randomized, double-blind, placebo-controlled study. Endocrinol Diabetes Metab. 2021 Jan 20;4(2):e00222. doi: 10.1002/edm2.222. eCollection 2021 Apr. PMID 33855222
- [Derived] Al-Sari N, Schmidt S, Suvitaival T, Kim M, Trost K, Ranjan AG, Christensen MB, Overgaard AJ, Pociot F, Norgaard K, Legido-Quigley C. Changes in the lipidome in type 1 diabetes following low carbohydrate diet: Post-hoc analysis of a randomized crossover trial. Endocrinol Diabetes Metab. 2021 Jan 4;4(2):e00213. doi: 10.1002/edm2.213. eCollection 2021 Apr. PMID 33855215

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Carbohydrate Diet: < 100 grams of carbohydrate per day
  Low carbohydrate diet
- High Carbohydrate Diet: > 250 grams of carbohydrate per day
  High carbohydrate diet
Period: First Intervention Period
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Period: Second Intervention Period
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Started | 7 (This is a cross-over study. Therefore starters does not necessarily equal completers of period 1.) | 5
Completed | 7 | 3
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Cohort: Baseline characteristics are for the whole study cohort, not for each of study arm of the cross-over study
Arm/Group | Study Cohort
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
body mass index [Median (Inter-Quartile Range); unit: kg/m*m] | 25 [23.7 to 26.4]
diabetes duration [Median (Inter-Quartile Range); unit: years] | 19 [13 to 32]
HbA1c [Median (Inter-Quartile Range); unit: mmol/mol] | 58 [55 to 60]
insulin pump use [Median (Inter-Quartile Range); unit: years] | 7 [5 to 11]
daily carbohydrate intake [Median (Inter-Quartile Range); unit: grams] | 145 [135 to 177]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent in Euglycemia
Description: Time spent with glucose values 4.0-10.0 mmol/l assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Percentage of time | 68.6 (8.9) | 65.3 (6.5)

2. Secondary Outcome: Mean Glucose
Description: Mean glucose value assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
mmol/l | 8.8 (0.7) | 8.9 (0.7)

3. Secondary Outcome: Standard Deviation of Glucose
Description: Standard deviation of glucose values assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
mmol/l | 2.9 (0.4) | 3.3 (0.4)

4. Secondary Outcome: Coefficient of Variation of Glucose
Description: Coefficient of variation of glucose values assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
percentage | 32.7 (3.2) | 37.5 (3.6)

5. Secondary Outcome: Mean Amplitude of Glycemic Excursions
Description: Mean amplitude of glycemic excursions (MAGE) assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Population: CGM data were collected, but the calculation of MAGE was not conducted. The analysis plan was changed as a result of changes in the guidelines for reporting of CGM-based measures. To calculate MAGE would require extensive work, and the results would be of no clinical relevance. Funding aquired for this project covers only clinically relevant analysis and ultimately, MAGE was not calculated due to lack of funding.
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time Spent in Hypoglycemia
Description: Percentage of time spent with glucose values ≤ 3.9 mmol/l assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Percentage of time | 1.9 (1.8) | 3.6 (2.1)

7. Secondary Outcome: Time Spent in Hyperglycemia
Description: Time spent with glucose values > 10.0 mmol/l assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Percentage of time | 29.5 (9.0) | 31.1 (7.3)

8. Secondary Outcome: Change in A1c
Description: Change in hemoglobin A1c
Time Frame: From baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 13 | 10
mmol/mol | 1 (1) | 1 (0)

9. Secondary Outcome: AUC Low
Description: Difference in area under the curve <4.0 mmol/l assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Population: CGM data were collected, but the calculation of AUC low was not conducted. The analysis plan was changed as a result of changes in the guidelines for reporting of CGM-based measures. To calculate AUC low would require extensive work, and the results would be of no clinical relevance. Funding aquired for this project covers only clinically relevant analysis and ultimately, AUC low was not calculated due to lack of funding.
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: AUC High
Description: Difference in area under the curve >10.0 mmol/l assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Population: CGM data were collected, but the calculation of AUC high was not conducted. The analysis plan was changed as a result of changes in the guidelines for reporting of CGM-based measures. To calculate AUC high would require extensive work, and the results would be of no clinical relevance. Funding aquired for this project covers only clinically relevant analysis and ultimately, AUC high was not calculated due to lack of funding.
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Post Breakfast Glucose Excursion
Description: Difference in post breakfast glucose excursion assessed by continuous glucose monitoring
Time Frame: 12 weeks - from baseline to end of study
Population: Data cannot be reported because the data collection method was invalid.
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Severe Hypoglycemia
Description: Number of severe hypoglycemia episodes (glucagon or intravenous glucose administration)
Time Frame: From baseline to 12 weeks
Measure: Number; unit: events
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 14
events | 0 | 0

13. Secondary Outcome: Total Daily Dose
Description: Total daily insulin dose
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Units of insulin | 33.6 (8.1) | 43.2 (11.0)

14. Secondary Outcome: Total Daily Basal Insulin 24 Hour
Description: Total daily basal insulin dose in the time range 00:00-24:00
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Units of insulin | 18.5 (5.4) | 17.3 (5.4)

15. Secondary Outcome: Total Nightime Basal Insulin
Description: Total nighttime basal insulin in the time range 00:00-06:00
Time Frame: From baseline to 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-08

16. Secondary Outcome: Total Daytime Basal Insulin
Description: Total daytime basal insulin in the time range 06:00-24:00
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

17. Secondary Outcome: Total Daily Bolus Insulin
Description: Difference in total daily bolus insulin
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
Units of insulin | 15.1 (4.4) | 25.9 (7.3)

18. Secondary Outcome: Blood Glucose Readings
Description: Number of blood glucose readings
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

19. Secondary Outcome: Carbohydrate Servings
Description: Number of daily carbohydrate servings (one serving ≥ 15 grams)
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

20. Secondary Outcome: Body Composition
Description: Change in fat mass (% of total body weight) assessed by Dual-energy X-ray Absorptiometry
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: percentage of total body weight
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 13 | 10
percentage of total body weight | -0.2 (0.6) | 1.0 (0.0)

21. Secondary Outcome: Weight
Description: Change in weight
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 13 | 10
kilogram | 1.9 (0.3) | 1.7 (1.6)

22. Secondary Outcome: Hip Circumference
Description: Change in hip circumference
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 13 | 10
centimeter | 5.2 (10.8) | 4.6 (0.4)

23. Secondary Outcome: Waist Circumference
Description: Change in waist circumference
Time Frame: From baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 13 | 10
centimeter | -1.9 (0.5) | 0.0 (1.8)

24. Secondary Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmHg | 4 (1) | 12 (5)

25. Secondary Outcome: Diastolic Blood Pressure
Description: Change in diastolic blood pressure
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmHg | 2 (4) | 7 (4)

26. Secondary Outcome: Heart Rate
Description: Change in heart rate
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
beats per minute | 3 (0) | 1 (1)

27. Secondary Outcome: Diabetes Treatment Satisfaction
Description: Change in Diabetes Treatment Satisfaction Questionnaire score. Score range: 0-36, with higher values representing higher degrees of treatment satisfaction.
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
units on a scale | 3.8 (2.7) | 4.9 (4.6)

28. Secondary Outcome: Hypoglycemia Fear
Description: Change in Hypoglycemia Fear Survey score. Score range: 0-52, with higher scores indicating higher degrees of fear of hypoglycemia.
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
units on a scale | 0 (0.9) | 2.5 (6.0)

29. Secondary Outcome: Cholesterol
Description: Change in total cholesterol
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.4 (0.0) | 0.2 (0.3)

30. Secondary Outcome: HDL
Description: Change in HDL
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.6 (0.0) | 0.03 (0.05)

31. Secondary Outcome: LDL
Description: Change in LDL
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.2 (0.0) | 0.2 (0.2)

32. Secondary Outcome: Triglycerides
Description: Change in triglycerides
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.0 (0.1) | 0.1 (0.0)

33. Secondary Outcome: Free Fatty Acids
Description: Change in free fatty acids
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

34. Secondary Outcome: Sodium
Description: Change in sodium
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0 (1) | 1 (1)

35. Secondary Outcome: Potassium
Description: Change in potassium
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.2 (0.0) | 0.1 (0.1)

36. Secondary Outcome: Creatinine
Description: Change in creatinine
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
micromol/l | 2 (1) | 2 (1)

37. Secondary Outcome: Urate
Description: Change in urate
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

38. Secondary Outcome: Albumin
Description: Change in albumin
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
g/l | 1 (1) | 0 (0)

39. Secondary Outcome: Hemoglobin
Description: Change in hemoglobin
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.3 (0.1) | 0.2 (0.0)

40. Secondary Outcome: Leucocytes
Description: Change in leucocytes
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: cells/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
cells/l | 0.1 (0.2) | 0.2 (0.1)

41. Secondary Outcome: Thrombocytes
Description: Change in thrombocytes
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: cells/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
cells/l | 17 (1) | 6 (10)

42. Secondary Outcome: Iron
Description: Change in iron
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
micromol/l | 2 (4) | 4 (0)

43. Secondary Outcome: Transferrin
Description: Change in transferrin
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

44. Secondary Outcome: Ferritin
Description: Change in ferritin
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

45. Secondary Outcome: Folate
Description: Change in folate
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
micromol/l | 0.5 (0.1) | 0.3 (0.9)

46. Secondary Outcome: Vitamin B-12
Description: Change in vitamin B-12
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
pmol/l | 18 (8) | 35 (10)

47. Secondary Outcome: Magnesium
Description: Change in magnesium
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.03 (0.00) | 0.02 (0.00)

48. Secondary Outcome: Zinc
Description: Change in zinc
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
micromol/l | 1 (1) | 0 (1)

49. Secondary Outcome: U-alb-crea Ratio
Description: Change in urine albumin-creatinine ratio
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mg/mmol | 1 (4) | 3 (1)

50. Secondary Outcome: Supar
Description: Change in Supar
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

51. Secondary Outcome: CRP
Description: Change in CRP
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

52. Secondary Outcome: IL-1
Description: Change in IL-1
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
pg/ml | 0.2 (0.3) | 0.9 (1.1)

53. Secondary Outcome: IL-6
Description: Change in IL-6
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
pg/ml | 1.8 (7.1) | 6.5 (4.3)

54. Secondary Outcome: IL-8
Description: Change in IL-8
Time Frame: 12 weeks - from baseline to end of study
Reporting Status: Not Posted, anticipated posting 2026-08

55. Secondary Outcome: TNF-alpha
Description: Change in TNF-alpha
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
pg/ml | 2.3 (3.0) | 2.8 (2.6)

56. Other Pre Specified Outcome: Carbohydrate Intake
Description: Daily carbohydrate intake assessed by insulin pump download
Time Frame: 12 weeks - from baseline to end of study
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 11
grams per day | 98 (11) | 246 (34)

57. Other Pre Specified Outcome: Ketones
Description: Morning blood ketone values obtained 7 times during the study period. A single value was calculated for each study participant based on an average of the 7 datapoints.
Time Frame: Spot test at week 0, 2, 4, 6, 8, 10 and 12
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 14 | 12
mmol/l | 0.2 (0.1) | 0.1 (0.0)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Low Carbohydrate Diet | High Carbohydrate Diet
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Carbohydrate Diet (N=14) | High Carbohydrate Diet (N=12)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02888691/Prot_SAP_000.pdf